CLINICAL TRIAL: NCT02387814
Title: A Single-Dose Pharmacokinetic Study of Abemaciclib (LY2835219) in Subjects With Varying Degrees of Hepatic Impairment
Brief Title: A Study of Abemaciclib in Participants With Varying Degrees of Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15538; I3Y-MC-JPBV (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Abemaciclib: Normal Hepatic Function (Experimental): Single dose of Abemaciclib administered orally on Day 1 to participants with normal hepatic function.
  Interventions: Drug: Abemaciclib
- Abemaciclib: Mild Hepatic Impairment (Experimental): Single dose of Abemaciclib administered orally on Day 1 to participants with mild hepatic impairment.
  Interventions: Drug: Abemaciclib
- Abemaciclib: Moderate Hepatic Impairment (Experimental): Single dose of Abemaciclib administered orally on Day 1 to participants with moderate hepatic impairment.
  Interventions: Drug: Abemaciclib
- Abemaciclib: Severe Hepatic Impairment (Experimental): Single dose of Abemaciclib administered orally on Day 1 to participants with severe hepatic impairment.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered Orally
  Other Names: LY2835219

SUMMARY:
The study involves a single dose of a study drug called abemaciclib taken by mouth. The purpose of this study will be to measure how much study drug gets into the blood stream and how long the body takes to get rid of it when given to participants with mild, moderate, or severe liver impairment compared to healthy participants. In addition, the tolerability of the study drug will be evaluated.

This study will last approximately 3 weeks for each participant, including check-in and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be of non-child-bearing potential
* Have a body mass index of 18 to 40 kilograms per square meter (kg/m²)

Exclusion Criteria:

* No history of cardiovascular, renal, respiratory, gastrointestinal, endocrine or hematological disorders
* Have known allergies to abemaciclib, related compounds, or any components of the formulation
* No human immunodeficiency virus (HIV) infection or antibodies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - DaVita Clinical Research, Lakewood, Colorado
  - Clinical Pharmacology of Miami (CPMI), Miami, Florida
  - Orlando Clinical Research Center (OCRC), Orlando, Florida
  - Indiana University - Digestive and Liver Diseases, Indianapolis, Indiana
  - DaVita Clinical Research, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Abemaciclib: Normal Hepatic Function: 200 milligrams (mg) abemaciclib administered once, orally, to participants with normal hepatic function.
- Abemaciclib: Mild Hepatic Impairment: 200 mg abemaciclib administered once, orally, to participants with mild hepatic impairment.
- Abemaciclib: Moderate Hepatic Impairment: 200 mg abemaciclib administered once, orally, to participants with moderate hepatic impairment.
- Abemaciclib: Severe Hepatic Impairment: 200 mg abemaciclib administered once, orally, to participants with severe hepatic impairment.
Period: Overall Study
Arm/Group | Abemaciclib: Normal Hepatic Function | Abemaciclib: Mild Hepatic Impairment | Abemaciclib: Moderate Hepatic Impairment | Abemaciclib: Severe Hepatic Impairment
Started | 10 | 9 | 10 | 6
Received Abemaciclib | 10 | 9 | 10 | 6
Completed | 10 | 9 | 10 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received abemaciclib.
Groups:
- Abemaciclib: Normal Hepatic Function: 200 mg abemaciclib administered once, orally, to participants with normal hepatic function.
- Total: Total of all reporting groups
Arm/Group | Abemaciclib: Normal Hepatic Function | Abemaciclib: Mild Hepatic Impairment | Abemaciclib: Moderate Hepatic Impairment | Abemaciclib: Severe Hepatic Impairment | Total
Number analyzed (Participants) | 10 | 9 | 10 | 6 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (4.8) | 56.6 (4.4) | 58.8 (5.5) | 53.2 (6.2) | 56.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 2 | 13
  Male | 5 | 6 | 7 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4 | 8
  Not Hispanic or Latino | 8 | 7 | 10 | 2 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 0 | 7
  White | 7 | 7 | 7 | 4 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 10 | 6 | 35

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Abemaciclib and Active Metabolites
Time Frame: Day 1: Predose, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72, 96, 120, 144, 168, and 192 Hours Postdose
Population: All participants who received abemaciclib and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Abemaciclib: Normal Hepatic Function | Abemaciclib: Mild Hepatic Impairment | Abemaciclib: Moderate Hepatic Impairment | Abemaciclib: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 9 | 10 | 6
nanograms per milliliter (ng/mL)
  Abemaciclib | 133 (63) | 109 (65) | 83.9 (47) | 156 (44)
  LSN2839567 | 31.2 (57) | 26.0 (31) | 13.6 (71) | 17.4 (45)
  LSN3106729: number analyzed (Participants) | 10 | 9 | 8 | 6
  LSN3106729 | 10.4 (47) | 6.24 (27) | 4.96 (90) | 2.70 (41)
  LSN3106726 | 55.3 (40) | 37.7 (35) | 19.2 (71) | 14.0 (27)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity(AUC[0-inf]) of Abemaciclib and Active Metabolites
Time Frame: Day 1: Predose, 1, 2, 3, 4, 6, 8, 10, 24, 48, 72, 96, 120, 144, 168, and 192 Hours Postdose
Population: All participants who received abemaciclib and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*h/mL)
Arm/Group | Abemaciclib: Normal Hepatic Function | Abemaciclib: Mild Hepatic Impairment | Abemaciclib: Moderate Hepatic Impairment | Abemaciclib: Severe Hepatic Impairment
Number analyzed (Participants) | 10 | 9 | 10 | 6
nanograms*hours/milliliter (ng*h/mL)
  Abemaciclib | 4460 (61) | 4280 (58) | 4940 (51) | 9310 (49)
  LSN2839567: number analyzed (Participants) | 10 | 9 | 10 | 5
  LSN2839567 | 1420 (40) | 1090 (34) | 921 (46) | 846 (33)
  LSN3106729: number analyzed (Participants) | 10 | 8 | 5 | 1
  LSN3106729 | 480 (55) | 257 (42) | 211 (251) | 35.3 (NA) — Due to lack of samples with quantifiable LSN3106729 concentrations, AUC(0-inf) could only be calculated for 1 participant. (Individual value: 35.3 ng*h/mL).
  LSN3106726 | 3120 (40) | 2200 (39) | 1570 (57) | 1170 (30)

ADVERSE EVENTS:
Arm/Group | Abemaciclib: Normal Hepatic Function | Abemaciclib: Mild Hepatic Impairment | Abemaciclib: Moderate Hepatic Impairment | Abemaciclib: Severe Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 4/10 | 6/9 | 7/10 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib: Normal Hepatic Function (N=10) | Abemaciclib: Mild Hepatic Impairment (N=9) | Abemaciclib: Moderate Hepatic Impairment (N=10) | Abemaciclib: Severe Hepatic Impairment (N=6)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib: Normal Hepatic Function (N=10) | Abemaciclib: Mild Hepatic Impairment (N=9) | Abemaciclib: Moderate Hepatic Impairment (N=10) | Abemaciclib: Severe Hepatic Impairment (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days